CLINICAL TRIAL: NCT02505867
Title: The Role of Sleep Disordered Breathing in Heart Failure Admissions
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funding
Sponsor: Rami Khayat (Other)
Collaborators: Philips Respironics (Industry)
Responsible Party: Sponsor-Investigator, Rami Khayat, Principal Investigator, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013H0228
Record Dates: First submitted 2015-07-21; First posted 2015-07-22 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Sleep Apnea Syndromes; Heart Failure
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Device - ASV Therapy (Experimental): Participants are provided with Adaptive Servo Ventilation (ASV) device during inpatient hospitalization or shortly after discharge.
  Interventions: Device: Adaptive Servo Ventilation
- Control (No Intervention): No device provided

INTERVENTIONS:
Device: Adaptive Servo Ventilation — Participants are provided with an Adaptive Servo Ventilation (ASV) device for targeted treatment of SDB during inpatient hospitalization or shortly after discharge.
  Other Names: Bipap AutoSV
  Arms: Device - ASV Therapy

SUMMARY:
The purpose of this study is to evaluate the effect of in-hospital diagnosis and treatment of sleep disordered breathing (SDB) on post-discharge mortality and readmissions in- hospitalized patients with acute heart failure syndrome and reduced ejection fraction (HFrEF).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effect of in-hospital diagnosis and treatment of sleep disordered breathing (SDB) on post-discharge mortality and readmissions in- hospitalized patients with heart failure and reduced ejection fraction (HFrEF). The study is a randomized controlled trial in HFrEF patients who are hospitalized with acute heart failure syndrome (AHFS) and have an in-hospital sleep study diagnostic of SDB. Participants will be randomized to either the current standard of care of AHFS treatment or an intervention arm in which expedited treatment with adaptive servo ventilation is initiated immediately upon in-hospital diagnosis of SDB.

ELIGIBILITY:
Inclusion Criteria:

1. Admission diagnosis of heart failure and AHFS as defined by the following: A chief complaint of dyspnea or fatigue; elevated left ventricular pressure. Elevated left ventricular pressure is indicated by at least one of the following: signs of volume overload pedal edema, crackles, consistent chest X-ray, increased measurement of left ventricular end-diastolic diameter or volume, or elevated BNP level.
2. Previously unrecognized or recognized but untreated SDB diagnosed or confirmed on attended inpatient sleep study during the index hospitalization with AHFS. SDB is defined as one of the following syndromes:

   1. AHI>15 with more than 50% apneas being central (CSA); or
   2. AHI>30 events with more than 50% of the events being obstructive (severe OSA) in patients with LVEF <30%.
3. Projected length of stay >2 days on admission day to ensure uniformity of the underlying severity of the AHFS and to enable the introduction of the ASV device and education
4. LVEF <45% within 1 year of admission. An echocardiogram may be performed to confirm the LVEF during the hospitalization to determine eligibility.
5. Ongoing targeted treatment for heart failure during the current hospitalization including at least one of the following: IV diuretics, IV infusion of inotropes or vasodilators, or planned revascularization, or device therapy.

Exclusion criteria:

1. Patients who were on supplemental oxygen for an indication other than SDB or heart failure prior to admission. These are patients who have chronic respiratory insufficiency.
2. Patients on treatment targeting CSA or OSA (ASV, oxygen, or CPAP); and patients who already provided and rejected positive airway pressure therapy due to intolerance of the pressure or the claustrophobia.
3. Cardiogenic shock and hemodynamic instability with MAP less than 55 mmHg off vasopressors, or concurrently on vasopressor treatment, left ventricular assist devices, or intra-aortic Balloon Pump. Inotropic agents will not constitute an exclusion criterion. Patients will be eligible once more stable off vasopressors.
4. Acute respiratory failure or insufficiency defined by (PaO2/FIO2) ratio less than 250, or FIO2 requirement more than 40%. Patients are eligible to participate once their FIO2 requirement is below 30%.
5. Overt neurological deficit or patients who arrived from a long-term care facility or expected to be discharged to one; and patients who have very poor functional outcome precluding ability to use the ASV device independently
6. Renal failure requiring renal replacement therapy; Patients will not be excluded if they were undergoing ultra-filtration for volume removal.
7. Moderate to severe chronic obstructive lung disease (FEV1/FVC < 55%).
8. Patients who are likely to receive heart transplant or left ventricular assist device (LVAD) in the subsequent year. These are patients who have high standing on the transplant list during the index hospitalization or have a cardiothoracic evaluation for implantation of LVAD.
9. Patients on long term or "bridging" inotropic infusion, or short life expectancy due to concomitant illness or heart failure
10. Patients who report severe sleepiness or who consider themselves at risk while driving.
11. Patients who fail the secondary screening procedure. Secondary screening procedure involves the patient being asked to wear the device and experience the pressure delivery for at least 30 minutes while relaxed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-11; Primary Completion 2016-12-01 (Actual); Study Completion 2016-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Khayat, MD, Principal Investigator — Ohio State University; William Abraham, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Device - ASV Therapy | Control
Started | 6 | 6
Completed | 0 | 0
Not Completed | 6 | 6
Not completed — Lack of Efficacy | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Device - ASV Therapy | Control | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Full Range); unit: years] | 47.33 [29 to 66] | 46.33 [31 to 72] | 46.83 [29 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Hospital Readmissions
Description: Number of participant hospital readmissions
Time Frame: Six Months
Measure: Count of Participants; unit: Participants
Arm/Group | Device - ASV Therapy | Control
Number analyzed (Participants) | 6 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Device - ASV Therapy | Control
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No